CLINICAL TRIAL: NCT01909635
Title: Assessment of Thoughts and Feelings Occurring During and After a Meal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision was made not to start the study before it was initiated.
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Dr. Hollie Raynor, Ph.D., R.D., The University of Tennessee, Knoxville
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 9230 B
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Behavior and Behavior Mechanisms; Food Habits; Feeding Behavior; Behavior
MeSH Terms: conditions — Behavior; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Food Feelings (Experimental): If you are randomized to this group, you will be asked to think about your feelings of hunger, fullness, and the sensory qualities of the food (such as texture, smell, flavor) as you eat your meal.
  Interventions: Behavioral: Food Feelings
- Other Feelings (Experimental): If you are randomized to this group, you will be asked to think about how hot or cold you feel, and how tired you are feeling as you eat your meal.
  Interventions: Behavioral: Other Feelings

INTERVENTIONS:
Behavioral: Food Feelings
  Arms: Food Feelings
Behavioral: Other Feelings
  Arms: Other Feelings

SUMMARY:
Kelsey Wallour and Dr. Hollie Raynor are doing a study to investigate the effect of focusing on certain thoughts and feelings during a meal on liking of items in the meal. A total of 36 women are anticipated to participate in this study.

DETAILED DESCRIPTION:
During the orientation, informed consent will be obtained, questionnaires about your thoughts and feelings will be completed, and height and weight will be measured to calculate BMI. Next, for the remaining eligible participants, both meal sessions will be scheduled within a two-week period, with the sessions scheduled within one hour of being at the same time of day. These sessions will be scheduled at dinnertime, between four pm and seven pm, with each session lasting approximately 75 minutes. Before leaving the orientation session, you will be instructed to not exercise on either of the days of the sessions. You will also be instructed to not eat four hours before either of your sessions, but to eat in a similar manner earlier in the day for each session.

You will be randomized to one of two groups in which you will be asked to think about different things during your meal.

Group 1: If you are randomized to this group, you will be asked to think about your feelings of hunger, fullness, and the sensory qualities of the food (such as texture, smell, flavor) as you eat your meal.

Group 2: If you are randomized to this group, you will be asked to think about how hot or cold you feel, and how tired you are feeling as you eat your meal.

At the start of each meal session, you will complete a food recall to record what you have consumed that day prior to the scheduled session. Also, a seven-day physical activity recall will be collected prior to beginning the meal. If you have not followed directions regarding eating and exercise, the session will be rescheduled.

Next you will rate your hunger, fullness, and liking of each food in the meal on a scale. Then you will be instructed to consume a bowl of chocolate pudding within five minutes. When you have completed the pudding, there will be a 30-minute rest period in which you will be allowed to read or study. After the rest period and before the meal begins, you will again rate on the scale your hunger, fullness, and liking of each food in the meal. Then you will be asked to silence or turn off any electronic devices, after which the researcher will facilitate a brief raisin eating exercise. After the raisin eating exercise, the researcher will bring in your meal. The meal will last for 30 minutes and will be videotaped, and you will eat until pleasantly full. At the end of the thirty minutes, the researcher will come in and remove the food and you will rate your feelings of hunger, fullness, and liking of the foods in the meal, and then you will be done with the session.

At the second session, the procedure will be exactly the same. In addition, you will complete several questionnaires about your thoughts and feelings after completion of the meal.

Please call Dr. Hollie Raynor at (865) 974-6259 if you have any questions about these procedures for the study.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-35 years old
* BMI greater than or equal to 25 kg/m2
* Unrestrained eater
* Do not have unfavorable preference or allergy to foods used in the investigation
* Do not have a health condition or use medication that affects eating or requires a therapeutic diet
* Must agree to instructions to not eat or exercise in stated hours before the sessions
* Must agree to come into HEAL for an orientation session, and two sessions where, each time, the participant will consume a preload followed by a thirty-minute ad libitum meal

Exclusion Criteria:

* Are pregnant or breastfeeding
* Are actively dieting to lose weight
* Report binge eating
* Do not meet one or more of the above mentioned eligibility requirements

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07 (Estimated); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Total grams of ad libitum meal consumed | 1 year
  The foods that will be used in this investigation are Tyson Chicken Breast Tenders, Ore-Ida Tater Tots, Birds Eye Steamfresh Pure & Simple green beans, and fresh oranges. Participants will be provided with ad libitum amounts of the foods, and the foods will be measured in grams to the tenth decimal point on an electronic food scale (Denver Instrument Co., Arvada, CO) before and after the meal. The weight of the container will also be measured. Total grams of each food consumed during the session will be determined by subtracting pre- and post-consumption weight of food.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, Ph.D., R.D., Principal Investigator — University of Tennessee; Kelsey Wallour, B.S.F.C.S., Principal Investigator — University of Tennessee
Locations (1):
- Healthy Eating and Activity Laboratory (HEAL), Knoxville, Tennessee, United States

REFERENCES:
- See also: Healthy and Activity Lab Information — http://heal.utk.edu/